CLINICAL TRIAL: NCT06726486
Title: Use of a Hypercaloric and Hyperprotein Supplement Enriched with Immunonutrients in Multi-pathological Malnourished Patients to Improve the Incidence and Prevalence of Pressure Sores: a Randomized Controlled Trial
Brief Title: Use of a Hypercaloric and Hyperprotein Supplement Enriched with Immunonutrients in Multi-pathological Malnourished Patients to Improve the Incidence and Prevalence of Pressure Sores
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Vegenat Healthcare (Unknown); Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Principal Investigator, Antonio Jesús Marín Paz, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84.21
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Multimorbidity; Comorbidity; Malnutrition; Pressure Ulcer Prevention
Keywords: Multimorbidity; Comorbidity; Malnutrition; Pressure Ulcer; Supplements; Immunonutrients
MeSH Terms: conditions — Malnutrition; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: A single-blind parallel Randomized Controlled Clinical Trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Atémpero) (Experimental): Participants received an arginine-enriched ONS called Atémpero®.
  Interventions: Dietary Supplement: Atémpero
- Control Group (Active Comparator): Participants received a complete high-protein, high-calorie diet with mixed fiber.
  Interventions: Dietary Supplement: Control (Standard treatment)

INTERVENTIONS:
Dietary Supplement: Atémpero — A complete hyperproteic and hypercaloric diet with a mixture of fibres enriched in omega 3, L-arginine and nucleotides (which provides vitamin C and Zinc) was administered.
  Arms: Intervention Group (Atémpero)
Dietary Supplement: Control (Standard treatment) — A complete high-protein and high-calorie diet with mixed fibre was administered.
  Arms: Control Group

SUMMARY:
The goal of this study is to evaluate the efficacy of a hypercaloric, hyperproteic enteral formula enriched with immunonutrients in preventing and treating pressure injuries in hospitalized malnourished patients.

Participants will take enteral formula (a complete hyperproteic and hypercaloric oral nutritional supplement with a fibre mixture enriched in omega 3, L-arginine and nucleotides, providing vitamin C and Zinc) or a hyperproteic and hypercaloric oral nutritional supplement with fibre mixture every day for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized chronic patients with complex needs in the Internal Medicine Department of a regional hospital.
* Malnourished or at risk of malnutrition.
* Moderate-high risk of developing pressure-related injuries or the presence of pressure-related injuries.

Exclusion Criteria:

* Limitations in oral intake (due to pathologies, state of health, among others).
* Contraindications for using the oral route and digestive intolerance or allergy to any of the components of the products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of pressure-related injuries | 15 and 30 days
  Dichotomous variable: Yes/No.
Risk of developing pressure-related injuries | 15 and 30 days
  Measurement instrument: Braden scale (low risk, moderate risk, high risk).
Categorization of pressure-related injuries | 15 and 30 days
  Measurement instrument: PUSH scale (I, II, III, IV).
Pressure-related injuries healing | 15 and 30 days
  Measurement instrument: PUSH scale (closed, epithelial tissue, granulation tissue, sphacelium, necrotic tissue).
Degree of dependence | 0, 15, and 30 days.
  Measurement instruments (description): Barthel score (independent, mild, moderate, severe).
Weight loss | 0, 15 and 30 days.
  Measurement instruments (description): Weight scale (kg).
% of dietary intake | 15 and 30 days.
  0%, 25%, 50%, 75%, 100% intake.
ONS adherence | 15 and 30 days.
  0%, 25%, 50%, 75%, 100% intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Punta Europa University of Cadiz, Algeciras, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Unending.
Access Criteria: All data from this study will be available upon request to the author by correspondence, under justified reasons.

REFERENCES:
- [Background] Liu P, Shen WQ, Chen HL. Efficacy of arginine-enriched enteral formulas for the healing of pressure ulcers: a systematic review. J Wound Care. 2017 Jun 2;26(6):319-323. doi: 10.12968/jowc.2017.26.6.319. PMID 28598762
- [Background] Barchitta M, Maugeri A, Favara G, Magnano San Lio R, Evola G, Agodi A, Basile G. Nutrition and Wound Healing: An Overview Focusing on the Beneficial Effects of Curcumin. Int J Mol Sci. 2019 Mar 5;20(5):1119. doi: 10.3390/ijms20051119. PMID 30841550
- [Background] Cheshmeh S, Hojati N, Mohammadi A, Rahmani N, Moradi S, Pasdar Y, Elahi N. The use of oral and enteral tube-fed arginine supplementation in pressure injury care: A systematic review and meta-analysis. Nurs Open. 2022 Nov;9(6):2552-2561. doi: 10.1002/nop2.974. Epub 2021 Jun 25. PMID 34170617
- [Background] Yatabe J, Saito F, Ishida I, Sato A, Hoshi M, Suzuki K, Kameda T, Ueno S, Yatabe MS, Watanabe T, Sanada H. Lower plasma arginine in enteral tube-fed patients with pressure ulcer and improved pressure ulcer healing after arginine supplementation by Arginaid Water. J Nutr Health Aging. 2011 Apr;15(4):282-6. doi: 10.1007/s12603-010-0306-4. PMID 21437560
- [Background] Roberts S, Chaboyer W, Desbrow B. Nutrition care-related practices and factors affecting nutritional intakes in hospital patients at risk of pressure ulcers. J Hum Nutr Diet. 2015 Aug;28(4):357-65. doi: 10.1111/jhn.12258. Epub 2014 Jun 27. PMID 24974729
- [Background] Eglseer D, Hodl M, Lohrmann C. Nutritional management of older hospitalised patients with pressure injuries. Int Wound J. 2019 Feb;16(1):226-232. doi: 10.1111/iwj.13016. Epub 2018 Nov 15. PMID 30440105
- [Background] Volkert D, Beck AM, Cederholm T, Cruz-Jentoft A, Hooper L, Kiesswetter E, Maggio M, Raynaud-Simon A, Sieber C, Sobotka L, van Asselt D, Wirth R, Bischoff SC. ESPEN practical guideline: Clinical nutrition and hydration in geriatrics. Clin Nutr. 2022 Apr;41(4):958-989. doi: 10.1016/j.clnu.2022.01.024. Epub 2022 Mar 5. PMID 35306388
- [Background] Langer G, Wan CS, Fink A, Schwingshackl L, Schoberer D. Nutritional interventions for preventing and treating pressure ulcers. Cochrane Database Syst Rev. 2024 Feb 12;2(2):CD003216. doi: 10.1002/14651858.CD003216.pub3. PMID 38345088
- [Background] Mervis JS, Phillips TJ. Pressure ulcers: Prevention and management. J Am Acad Dermatol. 2019 Oct;81(4):893-902. doi: 10.1016/j.jaad.2018.12.068. Epub 2019 Jan 18. PMID 30664906
- [Background] Banks MD, Ross LJ, Webster J, Mudge A, Stankiewicz M, Dwyer K, Coleman K, Campbell J. Pressure ulcer healing with an intensive nutrition intervention in an acute setting: a pilot randomised controlled trial. J Wound Care. 2016 Jul 2;25(7):384-92. doi: 10.12968/jowc.2016.25.7.384. PMID 27410392
- [Background] Clark RK, Stampas A, Kerr KW, Nelson JL, Sulo S, Leon-Novelo L, Ngan E, Pandya D. Evaluating the impact of using a wound-specific oral nutritional supplement to support wound healing in a rehabilitation setting. Int Wound J. 2023 Jan;20(1):145-154. doi: 10.1111/iwj.13849. Epub 2022 Jun 9. PMID 35684975
- [Background] Wood J, Brown B, Bartley A, Margarida Batista Custodio Cavaco A, Roberts AP, Santon K, Cook S. Reducing pressure ulcers across multiple care settings using a collaborative approach. BMJ Open Qual. 2019 Aug 20;8(3):e000409. doi: 10.1136/bmjoq-2018-000409. eCollection 2019. PMID 31523723
- [Background] Stracci G, Scarpellini E, Rinninella E, Mignini EV, Clementi N, Boni MV, Valeri MV, Sansoni D, Abenavoli L, Gasbarrini A, Rasetti C, Santori P. Effects of enteral nutrition on patients with pressure lesions: a single center, pilot study. Eur Rev Med Pharmacol Sci. 2020 Feb;24(3):1563-1570. doi: 10.26355/eurrev_202002_20214. PMID 32096205
- [Background] Wung Buh A, Mahmoud H, Chen W, McInnes MDF, Fergusson DA. Effects of implementing Pressure Ulcer Prevention Practice Guidelines (PUPPG) in the prevention of pressure ulcers among hospitalised elderly patients: a systematic review protocol. BMJ Open. 2021 Mar 12;11(3):e043042. doi: 10.1136/bmjopen-2020-043042. PMID 33712523
- [Background] Jaul E, Barron J, Rosenzweig JP, Menczel J. An overview of co-morbidities and the development of pressure ulcers among older adults. BMC Geriatr. 2018 Dec 11;18(1):305. doi: 10.1186/s12877-018-0997-7. PMID 30537947
- [Background] Jaul E, Menczel J. A comparative, descriptive study of systemic factors and survival in elderly patients with sacral pressure ulcers. Ostomy Wound Manage. 2015 Mar;61(3):20-6. PMID 25751847
- [Background] Guest JF, Ayoub N, McIlwraith T, Uchegbu I, Gerrish A, Weidlich D, Vowden K, Vowden P. Health economic burden that different wound types impose on the UK's National Health Service. Int Wound J. 2017 Apr;14(2):322-330. doi: 10.1111/iwj.12603. Epub 2016 May 26. PMID 27229943
- [Background] Li Z, Lin F, Thalib L, Chaboyer W. Global prevalence and incidence of pressure injuries in hospitalised adult patients: A systematic review and meta-analysis. Int J Nurs Stud. 2020 May;105:103546. doi: 10.1016/j.ijnurstu.2020.103546. Epub 2020 Jan 31. PMID 32113142
- [Background] Saghaleini SH, Dehghan K, Shadvar K, Sanaie S, Mahmoodpoor A, Ostadi Z. Pressure Ulcer and Nutrition. Indian J Crit Care Med. 2018 Apr;22(4):283-289. doi: 10.4103/ijccm.IJCCM_277_17. PMID 29743767
- [Background] Ledger L, Worsley P, Hope J, Schoonhoven L. Patient involvement in pressure ulcer prevention and adherence to prevention strategies: An integrative review. Int J Nurs Stud. 2020 Jan;101:103449. doi: 10.1016/j.ijnurstu.2019.103449. Epub 2019 Oct 14. PMID 31706155
- [Background] Cichosz SL, Voelsang AB, Tarnow L, Hasenkam JM, Fleischer J. Prediction of In-Hospital Pressure Ulcer Development. Adv Wound Care (New Rochelle). 2019 Jan 1;8(1):1-6. doi: 10.1089/wound.2018.0803. Epub 2019 Jan 5. PMID 30705784
- [Background] Cereda E, Neyens JCL, Caccialanza R, Rondanelli M, Schols JMGA. Efficacy of a Disease-Specific Nutritional Support for Pressure Ulcer Healing: A Systematic Review and Meta-Analysis. J Nutr Health Aging. 2017;21(6):655-661. doi: 10.1007/s12603-016-0822-y. PMID 28537329